CLINICAL TRIAL: NCT04817306
Title: A Prospective, Multicenter Study on Development and Validation of the Performance of a cfDNA Methylation-based Model for Early Cancer Detection (Pan-canceR Early DetectIon projeCT, PREDICT Study)
Brief Title: Pan-canceR Early DetectIon projeCT (PREDICT)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Guangzhou Burning Rock Dx Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: RSCD2020001
Record Dates: First submitted 2021-03-23; First posted 2021-03-26 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Cancer
Keywords: Cancer; Cell-free DNA (cfDNA) methylation; Early detection
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cancer Arm: Participants with new diagnosis of cancer, from whom blood samples will be collected
  Interventions: Device: Multi-cancer early detection test
- Benign Diseases Arm: Participants with benign diseases corresponding to the tumor types in the Cancer Arm, from whom blood samples will be collected
  Interventions: Device: Multi-cancer early detection test
- Non-tumor (Healthy) Arm: Participants without known presence of malignancies or benign diseases, from whom blood samples will be collected
  Interventions: Device: Multi-cancer early detection test

INTERVENTIONS:
Device: Multi-cancer early detection test — Blood collection and multi-cancer early detection testing

SUMMARY:
PREDICT is a prospective, multicenter study for the early detection of pan-cancer through cell-free DNA (cfDNA) methylation-based model, in which approximately 14,000 participants will be enrolled. The development and validation of the model will be conducted in participants with cancers or benign diseases, along with non-tumor (healthy) individuals through a two-stage approach. The sensitivity and specificity of the model in cancer early detection will be evaluated, and the accuracy of the identification for tissue of origin will be obtained.

ELIGIBILITY:
Inclusion Criteria for All the Participants:

* Ability to provide a written informed consent
* 40-75 years old

Exclusion Criteria for All the Participants:

* Inability to comply with study procedures
* Pregnancy or lactating women
* Recipients of organ transplant or prior non-autologous (allogeneic) bone marrow transplant or stem cell transplant
* Recipients of blood transfusion within 7 days prior to study blood draw
* Recipients of any anti-cancer therapy within 30 days prior to study blood draw, due to diseases other than cancer

Inclusion Criteria for Cancer Arm Participants:

* Confirmed diagnosis of a cancer or highly suspicious cases of cancer within 42 days prior to study blood draw. Tumor types in this study include lung cancer, colorectal cancer, liver cancer, ovarian cancer, gastric cancer, esophageal cancer, pancreatic cancer, biliary tract cancer, squamous cell carcinoma of the head and neck (except nasopharyngeal carcinoma)
* No prior or ongoing anti-cancer therapy (local or systematic) prior to study blood draw

Exclusion Criteria for Cancer Arm Participants:

* Known prior diagnosis of malignancies
* Other current malignant diseases or multiple primary tumors
* No confirmed diagnosis of cancer by histopathological or radiological assessments within 42 days of study blood draw, or diagnosis of a benign disease by histopathological assessments, or inability to characterize whether the lesion is malignant or benign
* Non-small-cell lung cancer patients with ground-class nodularity by radiological examination

Inclusion Criteria for Benign Diseases Arm Participants:

* Histopathologically confirmed or highly suspicious for benign diseases corresponding to the tumor types in the Cancer Arm within 90 days prior to study blood draw, or highly suspicious for benign diseases corresponding to the tumor types in Cancer Arm by radiological assessments or other clinical examinations
* No prior treatment of benign disease prior to study blood draw

Exclusion Criteria for Benign Diseases Arm Participants:

* Current or history of malignancies or precancerous lesions
* No confirmed diagnosis or inability to characterize a benign disease by radiological, endoscopic or histopathological assessments within 42 days of study blood draw

Inclusion Criteria for Non-tumor (Healthy) Arm Participants:

* No cancer-related symptoms or discomfort within 30 days prior to study blood draw
* No clinically significant finding by LDCT or abdominal ultrasound
* No clinically significant finding by breast ultrasound or Molybdenum Target Mammography Detection, or cervical liquid-based cell (TCT) detection for female participants
* No active hepatitis B or hepatitis C infection

Exclusion Criteria for Non-tumor (Healthy) Arm Participants:

* Prior or ongoing treatment of cancer within 3 years prior to study blood draw
* Unexplained weight loss
* Prior or current major diseases, including COPD, interstitial pneumonia, viral hepatitis, liver cirrhosis, inflammatory bowel disease
* Prior and current adenoma of the intestine and polyp of the intestine
* Changes in bowel habits, bowel abnormalities, hematochezia within 30 days prior to study blood draw
* Uncontrolled hypertension and other cardiovascular diseases
* Currently severe bleeding disorders
* Major surgery within 24 weeks prior to study blood draw
* Infection requiring anti-microbial therapy within 24 weeks prior to study blood draw
* Current autoimmunity disease
* Clinically significant or uncontrolled comorbidities which, in the investigator's opinion, should be excluded

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eligible participants will be recruited from medical centers and assigned into three arms, including participants with new diagnosis of cancer or corresponding benign diseases, and participants without the presence of malignancies or benign diseases.
Sampling Method: Non-Probability Sample
Enrollment: 14026 (Estimated)
Dates: Start 2021-03-29 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of early detection of cancer and Tissue of origin (TOO) accuracy of a cfDNA methylation-based model when specificity is 90%, 95% or 98% in healthy participants | 24 months
Sensitivity and specificity of early detection of cancer and TOO accuracy of a cfDNA methylation-based model | 24 months

SECONDARY OUTCOMES:
Sensitivity, specificity and TOO accuracy of a cfDNA methylation-based model in various types of cancer | 24 months
Sensitivity, specificity and TOO accuracy of a cfDNA methylation-based model in different stages of cancer | 24 months
Sensitivity, specificity and TOO accuracy of a cfDNA methylation-based model, in combination with clinical characteristics and other biomarkers | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Jia Fan, M.D., Ph.D, Principal Investigator — Shanghai Zhongshan Hospital
Locations (3):
- China (3):
  - Cancer Hospital, Chinese Academy of Medical Sciences & China National Cancer Center, Beijing, Beijing Municipality
  - Shanghai Ninth People's Hospital, Shanghai JiaoTong University, School of Medicine, Shanghai, Shanghai Municipality
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No